CLINICAL TRIAL: NCT05242718
Title: A Open Label, Multi-Dose, Multi-Period Exploratory Clinical Trial to Test Immune Diversity Response to Oral Dosing of Approved Nutritional Health Products at Approved Doses to Healthy Volunteers
Brief Title: Immune Diversity Response to Oral Dosing of Nutritional Health Products in Healthy Participants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Immunoflex Therapeutics Inc. (Industry)
Collaborators: Dicentra Inc. (Industry); University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMFX.CT1.002
Record Dates: First submitted 2022-01-13; First posted 2022-02-16 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Immunity Disorders
MeSH Terms: conditions — Immune System Diseases | interventions — Acetylcysteine; Echinacea extract; Curcumin; palmidrol

STUDY DESIGN:
Intervention Model Description: 8 participants assigned to Palmitoylethanolamide 8 participants assigned to Echinacea purpurea 8 participants assigned to Curcumin 8 participants assigned to N-Acetyl-L-cysteine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- N-Acetyl-L-cysteine (NAC) (Active Comparator): 600 mg 1 capsule twice daily for 14 days
  Interventions: Dietary Supplement: N-Acetyl-L-cysteine (NAC)
- Echinacea purpurea (Active Comparator): 252 mg 1 capsule twice daily for 14 days
  Interventions: Dietary Supplement: Echinacea purpurea
- Curcumin (Active Comparator): 60 mg 3 capsules once daily for 14 days
  Interventions: Dietary Supplement: Curcumin
- Palmitoylethanolamide (Active Comparator): 400 mg 3 capsules once daily for 14 days
  Interventions: Dietary Supplement: Palmitoylethanolamide

INTERVENTIONS:
Dietary Supplement: N-Acetyl-L-cysteine (NAC) — Health Canada Natural Product Number (NPN) 80056946
  Other Names: NAC
  Arms: N-Acetyl-L-cysteine (NAC)
Dietary Supplement: Echinacea purpurea — Health Canada Natural Product Number (NPN) 80093896
  Arms: Echinacea purpurea
Dietary Supplement: Curcumin — Health Canada Natural Product Number (NPN) 80043455
  Arms: Curcumin
Dietary Supplement: Palmitoylethanolamide — Health Canada Natural Product Number (NPN) 80097472
  Arms: Palmitoylethanolamide

SUMMARY:
A Phase IV, open-label, adaptive, 4-arm, multi-dose, single-centre, exploratory trial to assess the immune diversity response to oral administration of licensed Natural Health Products, in healthy adults, 60-70 years of age.

DETAILED DESCRIPTION:
In this study, the effect of licensed Natural Health Products (NHP) on immune response-related/antibody diversity parameters will be measured. Immune repertoire changes will be measured by genetic sequencing of segments of mRNA in the participant's blood that correspond to the coding regions for the Complementarity Determining Region - 3 (CDR-3) of T- and B-cell surface receptors. CDR-3 receptor segments are the highly variable recognition elements of the T- and B-cell receptors responsible for the recognition of foreign cells and other entities. This recognition step is an early step in the adaptive immune response.

Each of the four arms in the study contains 8 participants and each arm is assigned one NHP: Palmitoylethanolamide, or Echinacea purpurea, or Curcumin, or N-Acetyl-L-cysteine (NAC).

Longitudinal changes in immune diversity and dynamics, as indicated by changes in the CDR-3 sequence information will be measured over five timeframes in an four week period.

Baseline dynamics and diversity will be measured by comparing the results from participant visits 2 and 3. The impact of the NHP will be evident from comparing results between Visits 3 and 4. Finally, the impact of stopping the NHP dosing will be evident in comparing the results from Visit 5 to those of 4, 3, and 2. The techniques being used to analyze the sequence information are exploratory.

ELIGIBILITY:
Inclusion Criteria:

* Subjects meeting all of the following criteria will be considered for admission to the study:

  1. Healthy subjects between 60-70 years of age.
  2. Availability of the subject for one of the forecasted study periods and willingness of the subject to adhere to protocol requirements, as evidenced by a signed Informed Consent Form
  3. Have a BMI between18.5-29.9
  4. Agrees not to use any over the counter, prescription, health supplement or dietary supplement from screening until the end of the study period.
  5. Agrees to refrain from vaccinations throughout the study period.
  6. Able to maintain their current routine level of physical activities throughout the study period
  7. Willing and able to agree to the requirements and restrictions of this study (including but not limited to: not consuming more than 2 standard alcoholic beverages a day [A standard alcoholic beverage is defined as 12 ounces of beer, five (5) ounces of wine, or 1.5 ounces of liquor]), not consuming cannabis products of any type.
  8. In good health as determined by lack of clinically significant abnormalities in health assessments (history, physical examination, laboratory tests) performed at screening as judged by the physician.
  9. Women will be those without child bearing potential

Exclusion Criteria:

* Subjects meeting any of the following criteria will not be eligible for the study:

  1. Have a known sensitivity or allergy to any of the study products
  2. Self-reported smokers
  3. Receipt or use of an investigational product in another research study within 30 days prior to Baseline (Visit 2) or currently participating in another research study
  4. Receipt of a vaccination of any type within 60 days prior to the baseline visit.
  5. Difficulty with venipuncture and/or poor venous access
  6. Any major surgery within 1 year of study drug administration
  7. Anticipated major surgeries or major life events (major travel or change in lifestyle conditions) forecast to occur during the anticipated study periods
  8. Blood transfusion within 8 weeks of study drug administration
  9. Donation of blood or plasma to a blood bank or clinical study within 8 weeks of study drug administration
  10. Any clinically significant abnormalities in vital signs, as judged by the investigator.
  11. Hypertension or on blood pressure lowering medication
  12. Subjects with medical conditions that might interfere with participation in the study or interpretation of the study results. These include serious chronic diseases such as diabetes, neurologic or psychiatric disease (including any previous suicidal symptoms or suicide attempts), cardiovascular disease, gastrointestinal disease, pulmonary disease, cancer, autoimmune diseases, immunodeficiencies, hepatic or renal diseases.
  13. History of prior significant cardiovascular disease, coronary artery disease, cardiovascular surgery, significant valvular disease, heart failure, arrhythmias, sick sinus syndrome or stroke
  14. History of clinically significant cerebrovascular, metabolic, pulmonary, neurological, hematological, autoimmune, endocrine disorders, including individuals with Type I or Type II diabetes, or other clinically significant medical condition that, in the opinion of the Investigator, may preclude safe study participation
  15. History of immune disorder (such as HIV/AIDS), hepatitis B or hepatitis C, or positive immune disorder diagnosis
  16. History of alcohol or substance abuse in the 12 months prior to screening
  17. History of cannabis product use, including Cannabidiol (CBD), in the 3 months prior to screening
  18. Any other medical or social condition that, in the judgment of the investigator, would preclude provision of informed consent, make participation in the study unsafe, complicate interpretation of study outcome data or otherwise interfere with achieving the study objectives.

Ages: 60 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2021-01-10 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-20 (Actual)

PRIMARY OUTCOMES:
Change in participants T & B cell Diversity Index (D50) from day 0 to day 29 | 4 weeks
  D50 measures changes in frequency distributions of complementarity-determining region 3 (CDR3) in order to identify correlations between treatment and immune diversity. Diversity Index (D50) is a measure of the CDR3 diversity in the first half of the immune repertoire when looking at the frequency distributions. Additional bioinformatic analysis methods will be applied including Shannon Equitability Index and Antigen-specific Lymphocyte Identification by Clustering of Expanded Sequences.

CONTACTS AND LOCATIONS:
Overall Officials: Gurinder Raj, MD, Principal Investigator — dicentra
Locations (1):
- Dicentra, Toronto, Ontario, Canada